CLINICAL TRIAL: NCT04396574
Title: A Phase 3, 12-Month, Open-Label Study of Lasmiditan in Pediatric Patients With Migraine - PIONEER-PEDS2
Brief Title: A 12-Month Study of Lasmiditan (LY573144) Treatment in Children Aged 6 to 17 With Migraine
Acronym: PIONEER-PEDS2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16930; H8H-MC-LAHW (Other: Eli Lilly and Company); 2019-004379-38 (EudraCT Number)
Record Dates: First submitted 2020-05-18; First posted 2020-05-20 (Actual); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Migraine
Keywords: acute; long-term; open label; safety
MeSH Terms: conditions — Migraine Disorders | interventions — lasmiditan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lasmiditan Dose 1 (Experimental): Lasmiditan administered orally.
  Interventions: Drug: Lasmiditan
- Lasmiditan Dose 2 (Experimental): Lasmiditan administered orally.
  Interventions: Drug: Lasmiditan

INTERVENTIONS:
Drug: Lasmiditan — Administered orally
  Other Names: LY573144

SUMMARY:
The reason for this 12-month, open-label study is to see if the study drug lasmiditan is safe and effective for the intermittent acute treatment of migraine in children aged 6 to 17. The study will last about 12 months and may include up to 7 visits.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have completed study H8H-MC-LAHX (NCT03988088) or study H8H-MC-LAHV (NCT number to be determined)
* Participants must weigh at least 15 kilograms (kg)

Exclusion Criteria:

* Participants must not be pregnant or nursing
* Participants must not have any acute, serious, or unstable medical condition
* Participants must not be actively suicidal or at significant risk for suicide, in the opinion of the investigator

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1000 (Estimated)
Dates: Start 2020-06-30 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Treatment Emergent Adverse Events (TEAEs) by Treated Migraine Attack | Baseline through 12 Months
  Percentage of TEAEs by Treated Migraine Attack
Percentage of Participants with Discontinuations Due to Adverse Events (AEs) | Baseline through 12 Months
  Percentage of Participants with Discontinuations Due to AEs

SECONDARY OUTCOMES:
Percentage of Treated Attacks with Pain Freedom at 2 Hours | 12 Months
  Percentage of Treated Attacks with Pain Freedom at 2 Hours
Percentage of Treated Attacks with Pain Relief at 2 Hours | 12 Months
  Percentage of Treated Attacks with Pain Relief at 2 Hours
Percentage of Treated Attacks with MBS Freedom at 2 Hours | 12 Months
  Percentage of Treated Attacks with Most Bothersome Symptom (MBS) Freedom at 2 Hours

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (133):
- United States (71):
  - Central Research Associates, Birmingham, Alabama
  - Rehabilitation & Neurological Services, Huntsville, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Perseverance Research Center, Scottsdale, Arizona
  - Center for Neurosciences, Tucson, Arizona
  - Arkansas Children's, Little Rock, Arkansas
  - Core Healthcare Group, Cerritos, California
  - Miller Children's & Women's Hospital Long Beach, Long Beach, California
  - Sensa Health, Los Angeles, California
  - Orange County Research Institute - Ontario, Ontario, California
  - Yale University School of Medicine, New Haven, Connecticut
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Wolfson Children's Hospital, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc. dba CNS Healthcare, Jacksonville, Florida
  - Biotech Pharmaceutical Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Ezy Medical Research, Miami Lakes, Florida
  - Suncoast Clinical Research, Inc., New Port Richey, Florida
  - Avanza Medical Research Center, Pensacola, Florida
  - Clinical Research Center of Florida, Pompano Beach, Florida
  - USF Health, Tampa, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Palm Beach Neurology, West Palm Beach, Florida
  - Pediatric Neurology P.A., Winter Park, Florida
  - Meridian Clinical Research, LLC, Savannah, Georgia
  - Rophe Adult and Pediatric Medicine/SKYCRNG, Union City, Georgia
  - Hawaii Pacific Neuroscience, Honolulu, Hawaii
  - Medical Research Partners, Ammon, Idaho
  - Velocity Clinical Research, Boise, Meridian, Idaho
  - Chicago Headache Center and Research Institute, Chicago, Illinois
  - Chicago Headache Center and Research Institute - Naperville, Naperville, Illinois
  - Qualmedica Research, LLC, Evansville, Indiana
  - Fort Wayne Neurological Center - West, Fort Wayne, Indiana
  - Josephson Wallack Munshower Neurology, PC, Indianapolis, Indiana
  - Deaconess Clinic - Gateway Health Center, Newburgh, Indiana
  - Integrated Clinical Trial Services, Inc., West Des Moines, Iowa
  - Qualmedica Research, LLC, Bowling Green, Kentucky
  - University of Kentucky Chandler Medical Center, Lexington, Kentucky
  - Qualmedica Research, LLC, Owensboro, Kentucky
  - Children's Hospital New Orleans, New Orleans, Louisiana
  - Velocity Clinical Research - New Orleans, New Orleans, Louisiana
  - Pharmasite Research, Inc., Baltimore, Maryland
  - ActivMed Practices and Research, Methuen, Massachusetts
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Michigan State University, East Lansing, Michigan
  - Minneapolis Clinic of Neurology - Burnsville Office, Burnsville, Minnesota
  - SKY Integrative Medical Center/SKYCRNG, Ridgeland, Mississippi
  - Children's Mercy Hospital, Kansas City, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Rochester Clinical Research, Inc., Rochester, New York
  - Monroe Biomedical Research, Monroe, North Carolina
  - Accellacare - Piedmont, Statesville, North Carolina
  - Accellacare - Winston-Salem, Winston-Salem, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Headache Center of Hope, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Frontier Clinical Research, LLC, Scottdale, Pennsylvania
  - Frontier Clinical Research, LLC, Smithfield, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - ARC Clinical Research at Four Point, Austin, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Pain and Headache Centers of Texas, Houston, Texas
  - ClinPoint Trials, Waxahachie, Texas
  - Medical Research Partners - Logan, Logan, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Everett, Washington
  - Seattle Children's Hospital, Seattle, Washington
  - Seattle Women's: Health, Research, Gynecology, Seattle, Washington
  - Marshall Medical Center, Huntington, West Virginia
  - Frontier Clinical Research, Kingwood, West Virginia
- Belgium (2):
  - UZ Brussel, Brussels
  - Private Practice - Dr. Sava Simona, Saint-Nicolas
- France (4):
  - CHU d'Amiens-Picardie - Hôpital Sud, Amiens
  - Centre Hospitalier Universitaire Estaing, Clermont-Ferrand
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Hospitalier Général de Mont de Marsan - Hôpital Layné, Mont-de-Marsan
- Germany (2):
  - Private Practice - Dr. Irma Schöll, Bad Homburg
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau
- India (6):
  - Artemis hospital, Gurugram
  - Mangala Hospital & Mangala Kidney Foundation, Mangalore
  - Getwell Hospital and Research Institute, Nagpur
  - G.B. Pant Institute of Postgraduate Medical Education & Research, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Bhakti Vedanta Hospital and Research Institute, Thane
- Italy (5):
  - Ospedale San Paolo Bari, Bari
  - IRCCS Istituto Neurologico Carlo Besta, Milan
  - Universita degli Studi della Campania Luigi Vanvitelli, Napoli
  - Fondazione Istituto Neurologico C. Mondino, Pavia
  - Ospedale Pediatrico Bambino Gesù, Roma
- Japan (16):
  - Hiroshima City Hospital, Hiroshima
  - Tanaka Neurosurgery&Headache Clinic, Kagoshima
  - Nagaseki Headache Clinic, Kai
  - Hikita Pediatric clinic, Kiryū
  - Konan Hospital, Kobe
  - Umenotsuji Clinic, Kochi
  - Tatsuoka Neurology Clinic, Kyoto
  - Japanese Red Cross Kyoto Daiichi Hospital, Kyoto
  - Shinagawa Strings Clinic, Minato
  - Nishinomiya Municipal Central Hospital, Nishinomiya
  - Yamaguchi Clinic, Nishinomiya
  - Hyogo College of Medicine, Nishinomiya
  - Tominaga Hospital, Osaka
  - Sendai Headache and Neurology Clinic, Sendai
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Tokyo Headache Clinic, Tokyo
- Mexico (5):
  - Centro de Investigacion Medica Aguascalientes, Aguascalientes
  - Unidad de Investigación en Salud, Chihuahua City
  - AGNI Research and Assessment S.C., Cuernavaca
  - PanAmerican Clinical Research - Guadalajara, Guadalajara
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey
- Netherlands (2):
  - Canisius-Wilhelmina Ziekenhuis, Nijmegen
  - Isala, locatie Zwolle, Zwolle
- Puerto Rico (4):
  - Dr. Samuel Sanchez PSC, Caguas
  - Puerto Rico Health Institute, Dorado
  - Ponce Medical School Foundation Inc., Ponce
  - Wellness clinical Research Vega Baja, Vega Baja
- Romania (2):
  - Prof. Dr. Alexandru Obregia Psychiatry Hospital, Bucharest
  - Spitalul clinic de urgenta pentru copii Sf. Maria, Iași
- Russia (2):
  - Limited Liability Company University Clinic of headaches, Moscow
  - Sibneyromed Urban Neurological Center, Novosibirsk
- Spain (6):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitari Parc Tauli, Sabadell
  - Hospital Universitario Virgen Del Rocio, Seville
  - Hospital Clínico Universitario de Valladolid, Valladolid
- United Kingdom (6):
  - Royal Hospital for Sick Children, Glagow
  - James Paget University Hospital, Great Yarmouth
  - Re:Cognition Health - London, London
  - Great Ormond Street Hospital For Children NHS Foundation Trust, London
  - Queen's Medical Centre, Nottingham University Hospitals, Nottingham
  - Stepping Hill Hospital, Stockport

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A 12-Month Study of Lasmiditan (LY573144) Treatment in Children Aged 6 to 17 With Migraine (PIONEER-PEDS2) — https://trials.lillytrialguide.com/en-US/trial/F62T11Ido5SUiPl26NA8f